CLINICAL TRIAL: NCT02244658
Title: Recombinant Human Thrombopoietin (rhTPO) in Management of Chemotherapy-induced Thrombocytopenia in Acute Myelocytic Leukemia: a Multicenter Clinical Trial
Brief Title: Recombinant Human Thrombopoietin (rhTPO) in Management of Chemotherapy-induced Thrombocytopenia in Acute Myelocytic Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RhTPO-AML thrombocytopenia
Record Dates: First submitted 2014-09-13; First posted 2014-09-19 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-03

CONDITIONS: Antineoplastic Adverse Reaction; Thrombocytopenia; Acute Myelocytic Leukemia
Keywords: chemotherapy-induced thrombocytopenia; recombinant human thrombopoietin; acute myelocytic leukemia
MeSH Terms: conditions — Thrombocytopenia; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhTPO (Experimental): rhTPO 1.0 μg/kg·d subcutaneously for 7~14 consecutive days
  Interventions: Drug: rhTPO
- control (No Intervention): no thrombopoietic agents

INTERVENTIONS:
Drug: rhTPO — rhTPO 1.0 μg/kg·d subcutaneously for 7~14 consecutive days
  Other Names: TPIAO; S20050048/49 (SFDA, China)
  Arms: rhTPO

SUMMARY:
Chemotherapy-related myelosuppression usually occurs in AML patients, which induces severe thrombocytopenia and haemorrhage, a leading cause of death. This clinical trial aims at evaluating efficacy and safety of rhTPO in management of chemotherapy-induced thrombocytopenia in acute myelocytic leukemia.

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicentre, randomized controlled trial of 80 adults with chemotherapy-induced thrombocytopenia from 8 medical centers in China. AML patients with PLT count <30×10^9/L during the previous cycle of chemotherapy are randomized into two groups that one receives rhTPO at 1.0μg/kg·d subcutaneously for 7~14 consecutive days and the other receives no rhTPO or other thrombopoietic factor. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* AML patients with PLT count <30×10^9/L during the previous cycle of chemotherapy to minimize the risk of clinically significant bleeding.

Exclusion Criteria:

* allergic history to biological agents; history of thrombotic or hemorrhagic diseases; M3 or M7 subtype; pregnancy; hypertension; cardiovascular disease; diabetes; liver and kidney function impairment;

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response | 21 days since the first administration
  days that PLT count rebound to 30×10^9/L, 50×10^9/L and 100×10^9/L, respectively, from the minimal level after the very cycle of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China